CLINICAL TRIAL: NCT04275180
Title: Efficacy of Argatroban in Acute Ischemic Stroke With Early Neurological Deterioration
Brief Title: Efficacy Argatroban in Ischemic Stroke With Early Deterioration (EASE)
Acronym: EASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yan-2019-293
Record Dates: First submitted 2020-02-04; First posted 2020-02-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-02

CONDITIONS: Acute Progressive Ischemic Stroke
MeSH Terms: interventions — argatroban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Standard medical treatment, including routine antiplatelet, blood pressure control, statins to stabilize plaque, etc.
- Argatroban group (Experimental): Argatraban is used on the basis of standard medical treatment.
  Interventions: Drug: Argatroban

INTERVENTIONS:
Drug: Argatroban — Argatroban plus standard medical treatment
  Arms: Argatroban group

SUMMARY:
Acute ischemic stroke (AIS) has the characteristics of high morbidity, high mortality, high disability rate and high recurrence rate. Progressive cerebral infarction (PIS) is a subtype of AIS, accounting for 10% - 40%. Because of the gradual aggravation of neurological deficit symptoms, it has a higher rate of disability and death, which brings heavy mental and economic burden to families, society and the country.

The progress of acute cerebral infarction is generally within 6 hours to 1 week after the onset of the disease. At present, it is considered that thrombus prolongation is one of the important pathogenesis of PIS. Heparin can reduce the incidence of post-stroke embolism, but its benefits are offset by the risk of hemorrhage due to the high risk of hemorrhage. The 2013AHA guidelines in the United States do not recommend it as a routine anticoagulant therapy. Therefore, reducing the risk of bleeding is the key to the anticoagulation therapy of PIS.

Argatroban is a new thrombin inhibitor. Its mechanism of action is to bind and inactivate thrombin (factor Ⅱ a) directly.Compared with traditional anticoagulants, argatroban not only has the advantages of good anticoagulant effect and rapid onset, but also has high safety. Therefore, this study aims to verify the clinical efficacy of Argatroban in the treatment of PIS in a large population.

In this study, 628 patients are expected to be enrolled into the study group. The experimental group and the control group are selected by dynamic random method. Both groups are given standard medical treatment, including routine antiplatelet, blood pressure control, statins to stabilize plaque, etc. The control group is only given standard medical treatment. In the experimental group, Argatroban is used on the basis of standard medical treatment. Both groups are treated for 7 days, and the second-class prevention standard medical treatment is given from the 8th to the 90th day. The main outcome measure is the good prognosis rate at the third month after PIS. The good prognosis was defined as the modified Rankin Scale (mRS) ≤ 3.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) has the characteristics of high morbidity, high mortality, high disability rate and high recurrence rate. Progressive cerebral infarction (PIS) is a subtype of AIS, accounting for 10% - 40%. Because of the gradual aggravation of neurological deficit symptoms, it has a higher rate of disability and death, which brings heavy mental and economic burden to families, society and the country.

The progression of acute cerebral infarction is generally within 6 hours to 1 week after onset. At present, the guidelines recommend early intravenous thrombolysis and endovascular thrombectomy for patients with PIS. However, due to the limitation of time window, family economy and other factors, less than 5% of patients can really receive intravenous thrombolysis and endovascular therapy. Therefore, most of the patients with PIS are still treated with conventional antiplatelet aggregation therapy. At present, the pathogenesis of PIS has not been clear. The study considers that stroke progress is formed by a variety of risk factors and mechanisms, including poor collateral circulation, thrombus prolongation, stroke recurrence, brain edema, reocclusion of arteries, hemorrhagic transformation, etc. Thrombus prolongation is one of the important mechanisms. At present, there is a lack of effective treatment for PIS, including anticoagulation, antiplatelet and so on. Heparin is a commonly used anticoagulant. It is believed that heparin can reduce the risk of post-stroke embolism, but its benefits are offset by the risk of bleeding. The 2013AHA guidelines in the United States do not recommend it as a routine anticoagulant therapy. Therefore, reducing the risk of bleeding is the key to the anticoagulation therapy of PIS.

Argatroban is a new thrombin inhibitor. Its mechanism of action is reversible binding via thrombin catalytic site, independent of antithrombin level in vivo, and directly binding and inactivating thrombin (factor IIA). Argatroban has a strong inhibition on fibrin formation and platelet aggregation caused by thrombin, but does not inhibit other serine proteases such as trypsin, XA factor Fibrinolytic enzyme and kallikrein can effectively improve the hypercoagulability of patients. Compared with traditional anticoagulants, argatroban not only has the advantages of good anticoagulant effect and rapid onset, but also has high safety. According to a study in Japan, argatroban is superior to heparin in the treatment of cardiogenic stroke and has higher safety; a meta-analysis involving 14 small sample studies in China shows that argatroban can effectively improve the neurological deficit of PIS and improve the ability of daily life. In terms of safety, compared with the control group, argatroban treatment group has no increase in bleeding events. Therefore, this study aims to verify the clinical efficacy of argatroban in the treatment of PIS in a large population.

In this study, 628 patients are expected to be enrolled into the study group. The experimental group and the control group are selected by dynamic random method. Both groups are given standard medical treatment, including routine antiplatelet, blood pressure control, statins to stabilize plaque, etc. The control group is only given standard medical treatment. In the experimental group, Argatroban is used on the basis of standard medical treatment. Both groups are treated for 7 days, and the second-class prevention standard medical treatment is given from the 8th to the 90th day. The main outcome measure is the good prognosis rate at the third month after PIS. The good prognosis was defined as the modified Rankin Scale (mRS) ≤ 3. Secondary efficacy evaluation indexes: 1. The proportion of mRS ≤ 2 in the third month of PIS; 2. mRS score in the first and third months of PIS; 3. NIHSS score in the seventh, first and third months of PIS; 4. The rate of composite events in the first and third months of PIS, including cerebrovascular events, myocardial infarction, angina pectoris and systemic embolism; 5. Recent changes in living ability, Barthel Index in the first and third months. Safety evaluation indicators: symptomatic intracranial hemorrhage within 7 days after PIS; cerebral hemorrhage within 7 days after PIS; adverse reactions and events reported by researchers.

ELIGIBILITY:
Inclusion Criteria:

* AIS patients with typical symptoms and signs within 48h, including those who received intravenous thrombolysis for 24 hours.
* The neurologic function deteriorated from 6h to 48h after the onset of the disease, and the NIHSS score increased by ≥ 2 points;
* Sign informed consent.

Exclusion Criteria:

* The diagnosis was cardiogenic cerebral embolism;
* In the patients with large area cerebral infarction of anterior circulation, the focus area was larger than 2 / 3 of the area of cerebral hemisphere;
* Patients with NIHSS score ≥ 21;
* Patients with conversion of intracranial hemorrhage;
* Patients with tirofiban;
* Patients with blood pressure ≥ 180 / 110mmhg after treatment;
* There were severe heart, liver and kidney dysfunction, such as LVEF < 40%, serum AST and ALT increased to 3 times of the upper limit of normal, creatinine clearance < 30ml / min;
* Patients with hematological diseases and those with bleeding tendency;
* In the past 6 months, the patients had a history of severe gastrointestinal hemorrhage;
* Allergic to argatraban;
* Patients (such as those with mental and mental disorders) who are not suitable for the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a 3-month modified Rankin Scale (mRS) score≤ 3 | 3 months
  mRS 0-6, higher indicate worse outcome

SECONDARY OUTCOMES:
proportion of patients with a 3-month modified Rankin Scale (mRS) score≤ 2 | 3 months
  mRS 0-6, higher indicate worse outcome
mRS score in the third month of PIS | 3 months
  mRS 0-6, higher indicate worse outcome
National Institute of Health stroke scale(NIHSS) scores in the third months of PIS | 3 months
  NIHSS 0-42, higher indicate worse outcome
The rate of composite events in the third months of PIS, including cerebrovascular events, myocardial infarction, angina pectoris and systemic embolism | 3 months
  Complex events include cerebrovascular events, myocardial infarction, angina pectoris and systemic embolism.
Recent changes in living ability, Barthel Index in the third months | 3 months
  Barthel Index 0-100, higher indicate better outcome

OTHER OUTCOMES:
Symptomatic hemorrhage transformation within 7 days after PIS | 7 days
  Increase of National Institute of Health stroke scale(NIHSS) scores caused by intracranial hemorrhage confirmed by imaging ≥ 4 points.
Parenchymal hemorrhage within 7 days after PIS | 7 days
  parenchymal hematoma is assessed on MRI or CT according to the second European-Australasian acute stroke study (ECASS II).
Adverse reactions and events reported by researchers | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ze Xin Chen, Study Chair — 2nd affiliated hospital of Zhejiang University, School of Medicine
Locations (6):
- China (6):
  - Min Lou, Hangzhou, Zhejiang
  - People's Hospital of Anji, Anji
  - Jiaxing Second Hospital, Jiaxing
  - Ninghai First Hospital, Ninghai
  - Quzhou Kecheng People's Hospital, Quzhou
  - Tongxiang Diyi Renmin Hospital, Tongxiang

REFERENCES:
- [Derived] Zhang X, Zhong W, Xue R, Jin H, Gong X, Huang Y, Chen F, Chen M, Gu L, Ge Y, Ma X, Zhong B, Wang M, Hu H, Chen Z, Yan S, Chen Y, Wang X, Zhang X, Xu D, He Y, Lou M, Wang A, Zhang X, Ma L, Lu X, Wang J, Lou Q, Qian P, Xie G, Zhu X, He S, Hu J, Wen X, Liu Y, Wang Y, Fu J, Fan W, Liebeskind D, Yuan C, Lou M. Argatroban in Patients With Acute Ischemic Stroke With Early Neurological Deterioration: A Randomized Clinical Trial. JAMA Neurol. 2024 Feb 1;81(2):118-125. doi: 10.1001/jamaneurol.2023.5093. PMID 38190136